CLINICAL TRIAL: NCT00092378
Title: A Randomized, Double-Blind, Placebo- and Active-Comparator-Controlled, Parallel-Group Study of Rofecoxib and Diclofenac Sodium in the Treatment of Post-Bunionectomy Surgery Pain
Brief Title: A Study of Two Approved Drugs in the Treatment of Post-Bunionectomy Surgery Pain (0966-234)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0966-234; 2004_072
Record Dates: First submitted 2004-09-22; First posted 2004-09-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Pain
Keywords: Bunionectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0966, rofecoxib
Drug: Comparator: diclofenac sodium, placebo

SUMMARY:
This purpose of this study is to compare the safety and effectiveness of two approved drugs in the treatment of pain following bunionectomy surgery.

DETAILED DESCRIPTION:
The duration of treatment is 5 days for rofecoxib and 1 day for diclofenac sodium.

ELIGIBILITY:
Inclusion Criteria:

* Bunion removal

Exclusion Criteria:

* Any known allergies to the study design

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2003-09-01 (Actual); Primary Completion 2003-12-01 (Actual); Study Completion 2003-12-01 (Actual)

PRIMARY OUTCOMES:
Overall analgesic effect over 8 hours

SECONDARY OUTCOMES:
Time to onset of analgesic effect.
The use of supplemental analgesia on Days 2-3.
Peak analgesic effect on Day 1.
Overall safety and tolerability.
The analgesic effect on Days 2-3.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Desjardins PJ, Black PM, Daniels S, Bird SR, Fitzgerald BJ, Petruschke RA, Tershakovec A, Chang DJ. A randomized controlled study comparing rofecoxib, diclofenac sodium, and placebo in post-bunionectomy pain. Curr Med Res Opin. 2004 Oct;20(10):1523-37. doi: 10.1185/030079904X3069. PMID 15462686
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html